CLINICAL TRIAL: NCT05688189
Title: Initial Temperature Setting of High Flow Nasal Cannula in Critically Ill Patients: a Pragmatic Randomized Trial
Brief Title: Initial Temperature of High Flow Nasal Cannula
Acronym: BEST/2022
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 6385
Record Dates: First submitted 2022-12-28; First posted 2023-01-18 (Actual); Last update posted 2023-02-17 (Actual); Status verified 2023-01

CONDITIONS: Oxygen Therapy
Keywords: HFNC, Patient Comfort, Temperature

STUDY DESIGN:
Who Masked: Investigator
Masking Description: The principal investigator and the research nurse will be blinded to block size and number. The person responsible for data analysis will be provided an anonymized dataset, thus rendering him/her blinded to the type of treatment the patients received.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- 37 degree centigrade (Experimental): The 37°C arm implies the setting of the temperature immediately at 37°C.
  Interventions: Device: different starting temperature setting of HFNC
- 34-37 degree centigrade (Experimental): The 34-37°C arm implies the setting of the temperature at 34°C and after 15 minutes at 37°C.
  Interventions: Device: different starting temperature setting of HFNC
- 31-34-37 degree centigrade (Experimental): The 31-34-37°C arm implies setting the temperature initially at 31°C, after 15 minutes at 34°C and after another 15 minutes at 37°C.
  Interventions: Device: different starting temperature setting of HFNC

INTERVENTIONS:
Device: different starting temperature setting of HFNC — The humidification temperature will be set based on the enrollment arm (37°C vs 34-37°C vs 31-34-37°C)

SUMMARY:
In the literature there are no indication on which is the best setting of the humidification temperature at the start of treatment with high flow nasal cannula (HFNC) in intensive care unit (ICU). The primary objective of this study is to understand whether there is a difference between the approaches to the humidification temperature for initiating HFNC treatment based on the perceived comfort of ICU patients.

We hypothesize that a gradual increase in temperature (31-34-37°C or 34-37°C) could lead to a different comfort as compared to 37°C as initial starting setting.

The secondary aim is to assess the patient's dryness and humidity level of the nose.

DETAILED DESCRIPTION:
This is a single-center, parallel arm (1:1:1) interventional, non-pharmacological, pragmatic randomized trial. Adult patients who need HFNC treatment for clinical indication will be enrolled and receive a different initial temperature of humidification.

The treatment with HFNC will be carried out as it normally happens for clinical practice, that is the doctor will decide the oxygen concentration, from 21 to 100%, and the flow, from 30 to 60 liters / minute (usually 40-60 liters / minute), according to the patient's level of hypoxia. For the specific purpose of this study, the humidification temperature will be set by the nurse based on the enrollment arm (37°C vs 34-37°C vs 31-34-37°C) rather than by clinical decision. The 37°C arm implies the setting of the temperature immediately at 37°C. The 34-37°C arm implies the setting of the temperature at 34°C and after 15 minutes at 37°C. The 31-34-37°C arm implies setting the temperature initially at 31°C, after 15 minutes at 34°C and after another 15 minutes at 37°C. After 30 minutes at 37°C (target temperature), the patient will be asked to indicate his comfort level, using 5 score visual numerical scale (VNS) ranging from 1 (extreme discomfort) to 5 (best comfort) and the dyspnea level, using Borg scale ranging from 1 (no dyspnea) to 10 (extreme dyspnea). The level of dryness of the nose, HFNC settings and vital signs will also be recorded for each step.

The treatment with HFNC will be provided with the AIRVO 2 (trade mark) system (Fisher & Paykel Healthcare, New Zealand).

All study procedures will be performed at the ICU of the Fondazione IRCCS (Scientific Institute for Research, Hospitalization and Healthcare) Ca' Granda Ospedale Maggiore Policlinico.

ELIGIBILITY:
Inclusion Criteria:

* Patients need HFNC as per clinical indication
* Patients without ICU delirium (CAM ICU negative)

Exclusion Criteria:

* Patients unable to express informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2023-01-18 (Actual); Primary Completion 2023-02-06 (Actual); Study Completion 2023-02-15 (Actual)

PRIMARY OUTCOMES:
Patient comfort | 30 minutes
  Difference in comfort score among study arms at 37°C using visual numerical scale (VNS) ranging from 1 to 5

SECONDARY OUTCOMES:
Patient nose dryness | 30 minutes
  Difference in dryness score among study arms at 37°C using visual numerical scale (VNS) ranging from 1 to 5
Patient nose humidity | 30 minutes
  Difference in humidity score among study arms at 37°C using visual numerical scale (VNS) ranging from 1 to 5

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Galazzi, PhD, Principal Investigator — Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico
Locations (1):
- Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mauri T, Galazzi A, Binda F, Masciopinto L, Corcione N, Carlesso E, Lazzeri M, Spinelli E, Tubiolo D, Volta CA, Adamini I, Pesenti A, Grasselli G. Impact of flow and temperature on patient comfort during respiratory support by high-flow nasal cannula. Crit Care. 2018 May 9;22(1):120. doi: 10.1186/s13054-018-2039-4. PMID 29743098
- [Background] Rochwerg B, Einav S, Chaudhuri D, Mancebo J, Mauri T, Helviz Y, Goligher EC, Jaber S, Ricard JD, Rittayamai N, Roca O, Antonelli M, Maggiore SM, Demoule A, Hodgson CL, Mercat A, Wilcox ME, Granton D, Wang D, Azoulay E, Ouanes-Besbes L, Cinnella G, Rauseo M, Carvalho C, Dessap-Mekontso A, Fraser J, Frat JP, Gomersall C, Grasselli G, Hernandez G, Jog S, Pesenti A, Riviello ED, Slutsky AS, Stapleton RD, Talmor D, Thille AW, Brochard L, Burns KEA. The role for high flow nasal cannula as a respiratory support strategy in adults: a clinical practice guideline. Intensive Care Med. 2020 Dec;46(12):2226-2237. doi: 10.1007/s00134-020-06312-y. Epub 2020 Nov 17. PMID 33201321
- [Background] Chikata Y, Izawa M, Okuda N, Itagaki T, Nakataki E, Onodera M, Imanaka H, Nishimura M. Humidification performance of two high-flow nasal cannula devices: a bench study. Respir Care. 2014 Aug;59(8):1186-90. doi: 10.4187/respcare.02932. PMID 24368861
- [Derived] Galazzi A, Gambazza S, Binda F, Dossena C, Cislaghi A, Adamini I, Palese A, Grasselli G, Laquintana D. The starting temperature of high-flow nasal cannula and perceived comfort in critically ill patients: A pragmatic randomized controlled trial. Nurs Crit Care. 2024 Nov;29(6):1601-1609. doi: 10.1111/nicc.13159. Epub 2024 Sep 18. PMID 39293494